CLINICAL TRIAL: NCT03096171
Title: Flourishing App: An Evaluation With High School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Elisa Kozasa, PhD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HIAE_App Florescer_Alunos
Record Dates: First submitted 2017-03-24; First posted 2017-03-30 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Emotional Stress
Keywords: Stress; Well-being; Positive Psychology
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Behavioral: Flourishing App Program This intervention is based on relaxation, well-being promotion, meditation practices and positive psychology principles. The program is being evaluated in a classroom format into another project and was adapted for this project in the application format for mobile devices. It will last for 16 weeks, with trainings of 20 minutes, four times a week.
  No Intervention: Control App This group will observe their psychological and physical condition (levels of stress and well-being) during their daily activities and social interactions for 8 weeks. After the evaluations, this group will receive the intervention (Flourishing App Program) for more 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control App (No Intervention): Initially this control group will have access to a Control App and after 8 weeks this goup will receive the intervention (Flourishing App Program).
- Flourishing App Program (Experimental): This group will receive the intervention Flourishing App Program for 16 weeks.
  Interventions: Behavioral: Flourishing App Program

INTERVENTIONS:
Behavioral: Flourishing App Program — This intervention is based on relaxation, well-being promotion, meditation practices and positive psychology principles. The program is being evaluated in a classroom format into another project and was adapted for this project in the application format for mobile devices. It will last for 16 weeks, with trainings of 20 minutes, four times a week.
  Arms: Flourishing App Program

SUMMARY:
This protocol proposes a well-being program, delivered through an application for mobile devices, based on meditation and positive psychology principles such as human development, the improvement of virtues, quality of life and well-being. The investigators hypothesize that this program offered in mobile application may promote well-being and reduce stress related problems in the participants. Objectives: To evaluate the effectiveness of a well-being program delivered through an application for mobile devices in a sample of high school students. Methods: Sixty high school students will be recruited. The participants will be randomized in two groups of 30 participants each one, half of them in the control group (GC) and the other half to the intervention group (GI).

DETAILED DESCRIPTION:
Introduction: Some very successful stress management programs are based on the principle of Mindfulness. This protocol proposes a well-being program, delivered through an application for mobile devices, based on meditation and positive psychology principles such as human development, the improvement of virtues, quality of life and well-being. In the modern world, young people are connected to new technologies and the use of applications can be a fun way to learn how to cope with stress and promote well-being. In this sense, the investigators hypothesize that this program offered in mobile application can be considered an interesting alternative for high school students who want to reduce symptoms related to stress and also promote well-being. Objectives: To evaluate the effectiveness of a well-being program delivered through an application for mobile devices in a sample of high school students. Methods: Sixty high school students will be recruited. The participants will be randomized in two groups of 30 participants each one, half of them in the control group (GC) and the other half to the intervention group (GI). The GI will participate in the Flourishing App Program, for eight weeks, while the GC will have access to a Control App. Then, after the evaluations, the GC will receive the intervention (Flourishing App Program), while the first group will repeat the use of the Flourishing App Program. Questions will be applied to evaluate the levels of stress and well-being of participants before and after the program and before and after each training period.

ELIGIBILITY:
Inclusion Criteria:

* Complete elementary school

Exclusion Criteria:

-

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in subjective symptoms of stress in the last 30 days | baseline, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  Sliding scale for stress level from 0 to 100
Changes in subjective symptoms of well-being in the last 30 days | baseline, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  Sliding scale for well-being level from 0 to 100

SECONDARY OUTCOMES:
Changes in subjective symptoms of stress at the moment | four times a week, before and after the period of each class (20 min)
  Sliding scale for stress level from 0 to 100
Changes in subjective symptoms of well-being at the moment | four times a week, before and after the period of each class (20 min)
  Sliding scale for stress level from 0 to 100

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No